CLINICAL TRIAL: NCT05368532
Title: Novel Excitability Protocol to Identify Alteration of Voltage-gated Ion Channels
Brief Title: Excitability Protocol: Voltage-gated Ion Channels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Jenny Tigerholm, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-2020001-1
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Temperature — The temperature will be reduced for approximately one hour.

SUMMARY:
The purpose of subproject 1 is to evaluate the accuracy of a nerve excitability protocol in healthy subjects before testing the protocol in diabetic neuropathy patients. The nerve excitability protocol has been derived by computational modeling to identify abnormalities of three subtypes of ion voltage-gated channels. These three ion channels are all altered in animal models of diabetic neuropathy and, therefore, are likely candidates for generating the altered excitability in diabetic neuropathy patients. The hypothesis for subproject 1 is that due to the unique dynamics of each subtype of voltage-gated ion channels, it is possible to identify abnormal voltage-gated ion channel alterations by altering the shape of the electrical stimulation.

ELIGIBILITY:
Inclusion Criteria: Healthy men and women in the age 18-80 years who speak and understand English.

Exclusion Criteria:

* Pregnancy or breast feeding
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous and present neurologic, musculoskeletal or mental illnesses (e.g., epilepsy, neuropathy, fibromyalgia and depression)
* Skin diseases
* Past history of conditions possibly leading to neuropathy
* Inability to cooperate
* Current use of medications that may affect the study, e.g., analgesics
* Previous traumatic experience of an electrical accident
* Consumption of alcohol or painkillers within the last 24 hours
* Participation in other pain studies throughout the study period
* Patients with cardiac diseases (e.g., pacemaker).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-31 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Perception threshold for the excitability | Approximately 5 minutes to estimate.
  The perception threshold will be estimated for a set of electrical stimuli. The perception threshold is defined as the transcutaneous electrical current needed for the participant to perceive the stimulus. The electrode will be placed on the arm. The perception threshold will be estimated by the method of limits and the psi method.

SECONDARY OUTCOMES:
Sensation | Approximately 5 minutes to estimate.
  The investigator will ask the participant to rate the sensation of electrical stimulation by a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Tigerholm, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No